CLINICAL TRIAL: NCT02046044
Title: Comparing the Effects of Digoxin and Ivabradine on Mortality and Morbidity in Chronic Heart Failure With Reduced Ejection Fraction and Sinus Rhythm
Brief Title: Digoxin Versus Ivabradine in Heart Failure With Reduced Ejection Fraction
Acronym: DIVA-REF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Kurtulus Karauzum, Kurtulus Karauzum, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KK&DU-Iva-Dig2014
Record Dates: First submitted 2014-01-20; First posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Heart Failure
Keywords: Heart failure; Digoxin; Ivabradine
MeSH Terms: conditions — Heart Failure | interventions — Digoxin; Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ivabradine (Experimental): Ivabradine: initial dose of 5 mg b.id. dose up-titration to 7,5 mg b.id. in 2 weeks due to the heart rate and maintaining the last dose during 6 months.
  Interventions: Drug: Ivabradine
- Digoxin (Experimental): Digoxin: Digoxin 0,25 mg once a day 5 days per week during 6 months.
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Digoxin
  Arms: Digoxin
Drug: Ivabradine
  Arms: Ivabradine

SUMMARY:
Study hypothesis: Comparing the effect of digoxin and ivabradine in chronic heart failure patients with a left ventricular ejection of 35% or lower and sinus rhythm with heart rate 70 beats per minute or higher, and who are taking maximal dose of a beta blocker if tolerated.

DETAILED DESCRIPTION:
Selected patients have chronic heart failure with left ventricular systolic dysfunction and sinus rhythm. They take optimal medical therapy.

ELIGIBILITY:
1. Inclusion Criteria:

   * Left ventricular ejection fraction of 35% or lower (Ischaemic or non-ischaemic etiology)
   * Sinus rhythm with heart rate of 70 beats per minute or higher
   * Symptomatic heart failure with functional capacity of New York Heart Association class II, III, IV
2. Exclusion Criteria:

   * Chronic renal failure with glomerular filtration rate <30 ml/min
   * Atrial fibrillation
   * Pace maker rhythm
   * Advanced stage chronic obstructive lung disease
   * Comorbidity with expected survival below 1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Cardiac function and functional status and biochemical parameters | After 6 months
  Cardiac function (echocardiography): Systolic function (left ventricular ejection fraction) and diastolic function (Doppler E/A ratio, tissue Doppler e/e1 ratio, Doppler deceleration time of the E wave, left atrium volume index) Maximal oxygen consumption will be evaluated with cardiopulmonary exercise testing Changes in proBNP level (serum value) after treatment

SECONDARY OUTCOMES:
Cardiovascular mortality | Up to 6 months
  Death from cardiovascular reasons
All cause mortality | Up to 6 months
  Death from any cause.
Hospital admission for worsening heart failure | Up to 6 months
Heart rate and blood pressure | After 6 months
  Changes in heart rate and blood pressure.

OTHER OUTCOMES:
Hospitalization for a cardiovascular reason | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kurtulus Karauzum, MD, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)